CLINICAL TRIAL: NCT01461681
Title: A Randomized Controlled Trial for Patients With Heart Failure
Brief Title: Improving Care of Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11-06859
Record Dates: First submitted 2011-10-17; First posted 2011-10-28 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Depression; Pain; Dyspnea; Quality of Life
Keywords: Palliative care; Symptom management; Heart failure
MeSH Terms: conditions — Depression; Pain; Dyspnea; Heart Failure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Symptom Management Service for heart failure (Experimental): Subjects randomized to the SMS-HF group will receive a comprehensive PC consultation by the interdisciplinary PC team at each site consisting of a nurse practitioner, physician, social worker and chaplain with 6 months of follow up. All members of the PC team are experienced PC clinicians. The SMS-HF intervention is based on National Quality Forum preferred practices and the National Consensus Project guidelines for quality PC. The SMS-HF will include assessment and management of symptoms, particularly focused on depression, pain and dyspnea, and a discussion of goals of care.
  Interventions: Procedure: Symptom Management Service for Heart failure
- Usual cardiology care (No Intervention): The usual cardiology care group will receive usual care provided by the HF clinic. We will assess symptoms and QoL at enrollment and symptoms, QoL, satisfaction, advance care planning documentation, and resource utilization at follow up 6 months later.

INTERVENTIONS:
Procedure: Symptom Management Service for Heart failure — The symptom management service for heart failure (SMS-HF) will begin in the hospital where the patient will be seen daily until discharge and continue with at least 6 contacts over the next 6 months with the first outpatient contact occurring in person in the HF clinic within a month of discharge. Of the subsequent 5 monthly contacts, at least 2 will be in person with the remainder by telephone. Additional contacts between the SMS-HF team and patient will be scheduled as needed. Patients discharged to a site other than home will have monthly contacts by telephone until they are able to attend the clinic. We will assess changes in depression, pain, dyspnea, and quality of life from baseline to 6 month follow-up.
  Other Names: SMS-HF
  Arms: Symptom Management Service for heart failure

SUMMARY:
Heart failure (HF) affects more than 5 million Americans and is a major source of morbidity and mortality. Despite optimal management, over half of patients with HF suffer from pain, dyspnea, fatigue, and depression that diminish quality of life (QoL). HF care also exacts a huge financial toll with yearly costs of $35 billion. Although consensus guidelines call for providing palliative care (PC) to patients with HF to relieve suffering and improve QoL, few receive it. The overall aim of this project is to conduct a randomized controlled trial (RCT) to determine if an interdisciplinary PC intervention (Symptom Management Service-HF [SMS-HF]) provided concurrently with standard cardiology care improves symptoms, QoL and satisfaction, and reduces resource utilization in outpatients with Class II-IV HF compared to standard cardiology care alone. Subjects assigned to the SMS-HF group will receive a 6-month interdisciplinary PC intervention based on the investigators successful SMS model of outpatient PC for oncology patients and focused on assessment and management of physical, emotional, social, and spiritual distress and discussion of treatment preferences. Innovations of this study are that it will rigorously assess the impact of the SMS-HF on patient outcomes and on resource utilization, a key component to ensuring program sustainability. The investigators research team of PC and HF experts is recognized for its PC research and has a proven record of collaborating, conducting RCTs of PC interventions, and studying outpatients with HF. The environment at UCSF is highly supportive of innovative research and of sustaining programs with demonstrated improvements in patient outcomes and operational effectiveness. The overall goal is to use the results from this study to support an application to the NIH for a multi-center RCT of the SMS-HF and to study similar models of concurrent PC for patients with other serious illnesses.

ELIGIBILITY:
* HF as primary Dx or symptomatic/active HF
* During index hospitalization or within the prior 6 months
* Age > 18
* Admit from: hospital, skilled nursing, home
* Medicine, Cardiology, and Heart Failure Services
* Co-morbidities can include end-stage renal disease, metastatic cancer, ICU/CCU care patients if able to consent and complete survey
* English speaking

Exclusion Criteria:

* Non-English speaking
* Previous consult by Palliative Care Service
* Pulmonary HTN
* Right Heart Failure
* LVAD
* PCI or CABG patient within this admission
* AS with planned surgical intervention
* Pre/post heart transplant
* Pre/post organ transplant within this admission
* Dementia (unable to consent)
* Homeless
* Active drug user
* Hospice enrolled patient
* GeriTraCC patients
* Does not have a UCSF physician
* Lives outside of the SF Bay Area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Assess change in depression using the Center for Epidemiologic Studies Depression Scale (CES-D) | Outcome measures will be assessed through month 6 post baseline
  Outcome measures will be assessed at baseline, 3-months and 6-months The CES-D is a 20-item measure that includes items pertaining to a range of depressive symptoms. Each symptom is assessed 'in the past week' and recorded on a 4-point numeric scale (0= "rarely or none of the time" to 3= "most or all of the time") providing a composite score (range 0 - 60). A score of 16 or higher is generally used to denote the presence of significant depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Z Pantilat, MD, Principal Investigator — UCSF School of Medicine
Locations (2):
- United States (2):
  - UCSF Medical Center, San Francisco, California
  - University of California San Francisco Medical Center, San Francisco, California

REFERENCES:
- [Derived] O'Riordan DL, Rathfon MA, Joseph DM, Hawgood J, Rabow MW, Dracup KA, De Marco T, Pantilat SZ. Feasibility of Implementing a Palliative Care Intervention for People with Heart Failure: Learnings from a Pilot Randomized Clinical Trial. J Palliat Med. 2019 Dec;22(12):1583-1588. doi: 10.1089/jpm.2018.0633. Epub 2019 May 17. PMID 31099698